CLINICAL TRIAL: NCT03784508
Title: Identification of Biomarkers of Response After Bariatric Surgery in Morbidly Obese Patients
Acronym: PREDI-BAR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Principal Investigator, Andreea Ciudin, Head of the Morbid Obesity Unit and Clinical Trials Department, Hospital Universitari Vall d'Hebron Research Institute
Other Study IDs: PR(AG)320-2018
Record Dates: First submitted 2018-09-04; First posted 2018-12-24 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Morbid Obesity
Keywords: morbid obesity; bariatric surgery; psychological profile
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool samples Blood samples DNA from saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Bariatric surgery: 200 consecutive patients that will undergo bariatric surgery as a routinary procedure at our site

SUMMARY:
The prevalence of obesity in Spain is about 21.6%. The discouraging results provided by dietary treatment, together with the lack of funding for pharmacological treatment, have led to the progressive use of bariatric surgery (CB). Besides weight loss, CB associates a beneficial effect on metabolic comorbidities. However, 25-30% of operated patients present a weight response considered inappropriate, they do not resolve their comorbidities and/or present a weight-regain shortly after surgery. Therefore, predictive strategies are necessary to allow a correct selection of obese patients who are candidates for CB.

The main hypothesis of the study is that various factors such as psychopathological profile, body composition and metabolic alterations related to morbid obesity can influence the response to bariatric surgery.

DETAILED DESCRIPTION:
The investigators have designed a prospective study in which 200 consecutive patients from the outpatient clinic of the Morbidly Obesity Unit of the Vall d'Hebron Hospital will be included, meeting criteria for bariatric surgery (with BMI> 40 kg / m2 or BMI> 35 kg /m2 in the presence of comorbidities) and will undergo surgery in the investigator's center between September 2018 and September 2019. All patients will undergo (baseline, month, 6, 12 and 24 month): complete clinical history, analysis complete biochemistry, 2 blood samples will be extracted to study metabolomics, stool sample for microbiota study, bioimpedance for the study of body composition, determination of AGEs in the skin and lens, cognitive function assessment, retinal function assessment by microperimetry and they will be asked to complete several specific questionnaires for the evaluation of the psychopathological profile and the dietetic survey.

ELIGIBILITY:
Inclusion Criteria:

* Patients fulfilling criteria for bariatric surgery (BS).
* Signed informed consent fir the BS and the study.
* Previous accomplishment of the preoperative protocol for the BS at our site.
* undergo BS between September 2018 and December 2019
* Able to read and understand the specific questionnaires.

Exclusion Criteria:

* Any contraindication for the bariatric surgery.
* Impossibility to follow-up at our site (eg: patients from outside out community).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Consecutive patients that are attended at our outpatient clinic of the Morbid Obesity Unit of Vall Hebron University Hospital, that will undergo BS between September 2018 and December 2019.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
Evolution of the body mass index in morbidly obesity patients after bariatric surgery (BS). | 24month
  For the assessment of the evolution after bariatric surgery the investigators will use the body mass index parameter (BMI), calculated with the following formula: Body mass index (BMI) will be calculated as weight (kg)/height (m2).
  Changes in BMI, will be evaluated at 1, 6, 12 and 24 month after bariatric surgery.
Evolution of the excess of weight loss % (EWL%) after bariatric surgery. | 24 month
  - Excess of weight loss % (EWL%) will be calculated using the following formula: pre-bariatric surgery weight (kg)-visit weight (kg)/pre-bariatric surgery weight (kg)- ideal weight (for BMI 25) (kg) x 100%. Changes in EWL% will be evaluated at 1, 6, 12 and 24 month after bariatric surgery.
Evolution of the total weight loss after bariatric surgery | 24 month
  -Total weight loss (TWL) will be calculated as: pre-bariatric surgery weight (kg)- visit weight (kg). Changes in TWL will be evaluated at 1, 6, 12 and 24 month after bariatric surgery.

SECONDARY OUTCOMES:
Evaluation of the body composition scores before and after bariatric surgery by means of bioimpedanciometry. | 24 month
  All the patients will undergo before and after bariatric surgery (after 1,6, 12, and 24 month) the bioimpedance Bodystat QuadScan 4000 evaluation. The results are expressed in kg of free fatty mass and fatty mass. The change in Kg of the free fatty mass and fatty mass regarding the baseline will be evaluated.
Evaluation of the Advanced Glycation End products (AGEs) before and after bariatric surgery. | 24 month
  All the patients will undergo AGEs evaluation before, at 6, 12, 24 months after bariatric surgery (eye and skin using CLEARPATH DS-120 and microCAYA-AGEreader respectively). The presence of the AGEs is automatically calculated as standard deviation from the normal values for age and gender. The differences between the baseline value, at 6,12 and 24 month will be evaluated.
Evaluation of neuropsychological scores before and after bariatric surgery: eating attitudes | 24month
  Eating Attitudes Test (EAT) evaluates the possible eating disorders of the patients. The test will be used before, at 6, 12, and 24month after bariatric surgery and the scores will be compared. The investigators will search for correlations with the BMI, EWL% and TWL changes. The subjects will have to answer 40 items, each of it measured from 0 to 3, total score may range between 0 and 120. The accepted cut-off for diagnosis eating disorders is more than 20 for spanish population.
Evaluation of neuropsychological scores before and after bariatric surgery: Attention-Deficit Hyperactivity Disorder (ADHD) | 24month
  ADHD rating scale will be used before, at 6, 12, and 24month after bariatric surgery and the scores will be compared. The investigators will evaluate the existence of correlations with the BMI, EWL% and TWL changes. The scale ranges between 0-27 points, the highest the value, the higher de attention deficit and hyperactivity.
Evaluation of neuropsychological scores before and after bariatric surgery: Sheehan Disability Inventory (SDI). | 24 month
  Sheehan Disability Inventory (SDI) scale will be used before, at 6, 12, and 24month after bariatric surgery and the scores will be compared. The investigators will evaluate the existence of correlations with the BMI, EWL% and TWL changes. The Sheehan Disability Inventory evaluates the social fobia and the score ranges between 0-30. A score > 15 is considered pathological.
Evaluation of neuropsychological scores before and after bariatric surgery: Zuckerman-Kuhlman Personality Questionnaire (ZKPQ). | 24month
  ZKPQ personality evaluation will be used before, at 6, 12, and 24month after bariatric surgery and the scores will be compared. The investigators will evaluate the existence of correlations with the BMI, EWL% and TWL changes. ZKPQ is a quantitative scale which evaluates 6 personality dimensions: aggressivity (19 points), anxiety (19 points), impulsivity (17 points), activity (17 points), sociability (17 points). There is no clear cut-off for this test. In consequence, there will be evaluated only the changes after the bariatric surgery, compared with the baseline score. The higher the score the higher the personality disorder.
Evaluation of neuropsychological scores before and after bariatric surgery: COPE- stress management strategies. | 24month
  COPE test will be used before, at 6, 12, and 24month after bariatric surgery and the scores will be compared. The investigators will evaluate the existence of correlations with the BMI, EWL% and TWL changes. COPE is a quantitative scale which evaluates 15 strategies of stress coping. The total score ranges between 15-60 points. There is a direct relation between the score and the ability to manage the stress, but no clear cut-off for this test exists. In consequence, we will only evaluate the changes after the bariatric surgery regarding the baseline score. The highest score indicates better strategies to cope the stress.
Evaluation of neuropsychological scores before and after bariatric surgery: ROTTER´s locus of control scale. | 24month
  ROTTER´s locus of control scale test will be used before, at 6, 12, and 24month after bariatric surgery and the scores will be compared. The investigators will evaluate the existence of correlations with the BMI, EWL% and TWL changes. COPE is a quantitative scale which a total score ranging between 0-29 points. The cut-off value <15 defines the internal locus of control.
Evaluation of neuropsychological scores before and after bariatric surgery: YALE food addiction. | 24month
  YALE food addiction scale test will be used before, at 6, 12, and 24month after bariatric surgery and the scores will be compared. The investigators will evaluate the existence of correlations with the BMI, EWL% and TWL changes. There is a direct relation between the score and the food addiction, is a quantitative scale but there is no clear cut-off. There will be evaluated the changes in the score at 6,12, and 24 month after the bariatric surgery, comparing with baseline. The highest the score, the higher the food addiction.
Evaluation of neuropsychological scores before and after bariatric surgery:The Bariatric Analysis and Reporting Outcome System (B.A.R.OS). | 24month
  B.A.R.O.S test will be used before, at 6, 12, and 24month after bariatric surgery and the scores will be compared. The investigators will evaluate the existence of correlations with the BMI, EWL% and TWL changes. B.A.R.O.S. is a quantitative questionnaire evaluating the quality of life after the bariatric surgery. The scale ranges between 0 and 9. The higher the score the highest the quality of life of the patient.
Evaluation of neuropsychological scores before and after bariatric surgery: The State-Trait Anxiety Inventory (STAI). | 24month
  STAI anxiety questionnaire evaluates the degree of the anxiety of the patient and will be used before, at 6, 12, and 24month after bariatric surgery and the scores will be compared. The investigators will evaluate the existence of correlations with the BMI, EWL% and TWL changes. The score ranges between 0 and 60. A cut-off value> 19 is considered pathological anxiety.
Evaluation of neuropsychological scores before and after bariatric surgery: WPAI (working productivity questionnaire). | 24month
  WPAI questionnaire will be used before, at 6, 12, and 24month after bariatric surgery and the results will be compared. The investigators will evaluate the existence of correlations with the BMI, EWL% and TWL changes. There is a qualitative score, evaluating the working status of the patient: retiree, active, off-work>6month, unemployed, permanent occupational disability. Percentages of each category will be evaluated at each time. Ej: % of unemployed, etc.
Evaluation of neuropsychological scores before and after bariatric surgery: Beck Depression Inventory (BDI) | 24month
  BDI evaluates if depression exists and its degree. It will be used before, at 6, 12, and 24month after bariatric surgery and the results will be compared. The investigators will evaluate the existence of correlations with the BMI, EWL% and TWL changes. The score ranges between 0-40. 0-10: normal; 10-16 mild emotional; 17-20: borderline clinical depression; 21-30 moderate depression; 31-40 severe depression.
Evaluation of the congnitive function before and after bariatric surgery | 24 month
  Minimental State Evaluation Test and Montreal Cognitive Assessment test will be used before and at 12 and 24 month after bariatric surgery
Evaluation of the utility of the retinal function evaluation in the detection of cognitive disfunction before and after bariatric surgery | 24 month
  Retinal microperimetry using MAIA 3rd generation microperimeter will be used before and at 12 and 24 month after the bariatric surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Andreea Ciudin, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No